CLINICAL TRIAL: NCT00808314
Title: Lexiscan(TM) Rb-82 Myocardial Perfusion Positron Emission Computed Tomography: A Comparison With Dipyridamole
Brief Title: Lexiscan(TM) Rb-82 Myocardial Perfusion PET: A Comparison With Dipyridamole Stress
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiovascular Imaging Technologies (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Timothy M. Bateman, MD, Principal Investigator, Cardiovascular Imaging Technologies
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-271
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Lexiscan(TM); Dipyridamole; Myocardial Perfusion; Positron Emission Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LL for CAD (Active Comparator): Subjects with <5% pre-test low likelihood for CAD based on Diamond and Forrester criteria will be recruited to undergo both rest/stress dipyridamole PET followed by a rest/stress Lexiscan(TM) PET with 30 days.
  Interventions: Drug: Rest/Dipyridamole Stress Rb-82 Myocardial Perfusion PET/CT; Drug: Rest/Lexiscan(TM) Stress Rb-82 Myocardial Perfusion PET
- CAD (Active Comparator): Subjects with existing mild-moderate ishemia demonstrated by a recent (< 1 month) rest/stress dipyridamole PET will undergo a rest/stress Lexiscan(TM) PET.
  Interventions: Drug: Rest/Lexiscan(TM) Stress Rb-82 Myocardial Perfusion PET

INTERVENTIONS:
Drug: Rest/Dipyridamole Stress Rb-82 Myocardial Perfusion PET/CT — A CT scan will be acquired for attenuation correction of the rest image (9 mA, 120 kVp, 4.24 secs) during end-expiration breath-holding. This will be followed by infusion of approximately 60 mCi of Rb-82, 60 to 100 seconds after which resting images will be acquired with ECG-gating. Following rest imaging, 0.56 mg/kg of dipyridamole will be infused over 4 minutes. Three minutes after the completion of the infusion, approximately 60 mCi of Rb-82 will be infused. Peak stress images will be acquired with ECG-gating, starting 90 seconds after the the beginning of the infusion of Rb-82 and continuing for 5 minutes. A CT scan will be acquired for attenuation correction of the stress image (9 mA, 120 kVp, 4.24 secs) during end-expiration breath-holding.
  Arms: LL for CAD
Drug: Rest/Lexiscan(TM) Stress Rb-82 Myocardial Perfusion PET — A CT scan will be acquired for attenuation correction of the rest image (9 mA, 120 kVp, 4.24 secs) during end-expiration breath-holding. This will be followed by infusion of approximately 60 mCi of Rb-82, 60 to 100 seconds after which resting images will be acquired with ECG-gating. Following rest imaging, 400 umg of Lexiscan(TM) will be injected, and then approximately 60 mCi of Rb-82 waill be infused. Peak stress images will be acquired in list mode with ECG-gating, starting 90 seconds after the the beginning of the infusion of Rb-82 and continuing for 5 minutes. A CT scan willbe acquired for attenuation correction of the stress image (9 mA, 120 kVp, 4.24 secs) during end-expiration breath-holding.

SUMMARY:
Lexiscan(TM) has ideal properties for Rb-82 PET imaging and the stress response it invokes may offer multiple advantages for the diagnosis of coronary disease and functional abnormalities. The goal of this investigation is to establish quantitative equivalence of Lexiscan(TM) rest/stress Rb-82 PET images to dipyridamole rest/stress images.

ELIGIBILITY:
Inclusion Criteria:

* BMI <35
* No intervention or change in management between dipyridamole and Lexiscan(TM) PET

Exclusion Criteria:

* BMI >35
* An intervention or change in management between dipyridamole and Lexiscan(TM) PET

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Quantitative analysis of local and regional myocardial perfusion between Lexiscan(TM) and dipyridamole rest/stress Rb82 PET | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Bateman, MD, Principal Investigator — Cardiovascular Imaging Technologies
Locations (1):
- Saint Luke's Cardiovascular Consultants, Kansas City, Missouri, United States